CLINICAL TRIAL: NCT07379242
Title: Lung Recruitment Assessed by Two-Dimensional/Three-Dimensional Electrical Impedance Tomography and Recruitment-to-Inflation Ratio in Acute Respiratory Failure Patients With Mechanical Ventilation
Brief Title: Lung Recruitment Assessed by 2D/3D-EIT and R/I Ratio in Acute Respiratory Failure Patients With Mechanical Ventilation
Status: Recruiting | Type: Observational
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 3D EIT-based PEEP & R/I ratio
Record Dates: First submitted 2026-01-21; First posted 2026-01-30 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Acute Respiratory Failure (ARF)
Keywords: Acute respiratory failure; PEEP titration; 3D-EIT; 2D-EIT; Lung recruitability; R/I ratio

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Mechanically ventilated patients with hypoxemia requiring clinical PEEP optimization: The study will enroll mechanically ventilated patients under sedation/analgesia without spontaneous breathing, exhibiting a oxygenation index (PaO₂/FiO₂ ratio) <300 mmHg, and deemed clinically eligible for PEEP titration by attending physicians.
  Interventions: Diagnostic Test: The lung recruitment potential assessed and PEEP titration by ventilator and 2D/3D EIT

INTERVENTIONS:
Diagnostic Test: The lung recruitment potential assessed and PEEP titration by ventilator and 2D/3D EIT — The patient will undergo a standardized PEEP titration procedure and determination of the Recruitment-to-Inflation ratio (R/I ratio), with concurrent monitoring by both 2D- and 3D- EIT.

SUMMARY:
The purpose of this observational study is to assess the differences and consistency in evaluating lung recruitment potential between the recruitment-to-inflation ratio (R/I ratio) and three-dimensional electrical impedance tomography (3D-EIT) and two-dimensional EIT (2D-EIT) in mechanically ventilated patients with acute respiratory failure. The main questions it aims to answer is:

Are the lung recruitment potentials predicted by 3D-EIT, 2D-EIT and the R/I ratio consistent? Participants will: Undergo a standardized PEEP titration protocol with synchronized EIT monitoring; Have R/I ratios measured at high and low PEEP levels.

ELIGIBILITY:
Inclusion Criteria:

* Mechanically ventilated patients under sedation and analgesia with no spontaneous breathing.
* Oxygenation index < 300 mmHg.
* Patients who are clinically judged by the attending doctor to require the PEEP titration.

Exclusion Criteria:

* Aged under 18 years.
* Pregnancy.
* Contraindications for EIT examination (e.g. automatic implantable cardioverter defibrillator, implantable pumps, chest wounds limiting electrode belt placement, severe thoracic deformity, and others).
* No informed consent obtained.
* Hemodynamic instability with intolerance to high PEEP levels determined by the attending doctor.
* High-risk populations with pneumothorax, mediastinal emphysema, and other such conditions determined by the attending doctor.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with acute respiratory failure who are intubated, under sedation and analgesia with controlled ventilation and no spontaneous breathing will be recruited from the Department of Critical Care Medicine, Peking Union Medical College Hospital. Additional inclusion criteria include an oxygenation index of less than 300 mmHg, clinical judgment indicating the need for PEEP titration, and no contraindications to PEEP titration or EIT examination.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2025-09-01 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Lung recruitment assessed by R/I ratio and 2D/3D-EIT （PEEP titration） | Within 24 hours post-enrollment
  Lung recruitment potential can be predicted by the R/I ratio and the lung collapse rate calculated from 2D/3D-EIT.

OTHER OUTCOMES:
R/I ratio measured by 2D/3D-EIT | Within 24 hours after enrollment
  The R/I ratio can be calculated from 2D/3D-EIT.
V/Q monitored by EIT | Within 24 hours after enrollment
  Ventilation and perfusion monitored by 2D/3D-EIT at different PEEP levels. To evaluate the V/Q match, deadspace and shunt lung region.
SpO₂ at different PEEP levels | Within 24 hours after enrollment
  Pulse oxygen saturation at different PEEP levels
Lung compliance at different PEEP levels | Within 24 hours after enrollment
  Lung compliance at different PEEP levels measured via ventilator parameters
Mechanical power | Within 24 hours after enrollment
  Mechanical power measured via ventilator parameters

CONTACTS AND LOCATIONS:
Overall Officials: Huaiwu He, Study Chair — Peking Union Medical College Hospital
Locations (1):
- Department of Critical Care Medicine, Peking Union Medical College Hospital, Peking Union Medical College, Chinese Academy of Medical Sciences, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No